CLINICAL TRIAL: NCT02594657
Title: Pedal Rate Influence on Oxygen Consumption in Eccentric
Acronym: PRIOx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: CHU-0241
Record Dates: First submitted 2015-07-09; First posted 2015-11-03 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: Eccentric; Ergometer; Pedal rate; Oxygen consumption; Only health volunteers

ARMS (2):
- pedal rate ON 50 RPM (Experimental)
  Interventions: Procedure: pedal rate on 50 RPM
- pedal rate on 80 RPM (Experimental)
  Interventions: Procedure: pedal rate on 80 RPM

INTERVENTIONS:
Procedure: pedal rate on 50 RPM — All measurements are performed in two pedalling situations. The two frequencies used will be 50 and 80 RPM. For each subject the running order (50 and 80, 80 and 50) is randomly determined
  Arms: pedal rate ON 50 RPM
Procedure: pedal rate on 80 RPM — All measurements are performed in two pedalling situations. The two frequencies used will be 50 and 80 RPM. For each subject the running order (50 and 80, 80 and 50) is randomly determined
  Arms: pedal rate on 80 RPM

SUMMARY:
Nowadays, ECC exercise can be realized using various modalities that target small or large muscle masses in a segmentary or dynamic way. The training program proposed in this study is realised on an handmade ergocycle which allows eccentric contractions.

With this type of ergometer, O2 consumption (VO2) is three to five fold lower than during an exercise realised at the same power output with a concentric ergocycle. Due to this later propertie, which origins are not yet fully identified, there is an increasing interest to embed ECC in rehabilitation programs.

The investigators hypothesis that a higher pedal rate will induce a lower oxygen consumption, with the same benefits.

This study aims to compare oxygen consumption at two pedal rates : 50 and 80 rotation per minute (rpm).

The ultimate goal is to assess efficacy and tolerance of eccentric training on ergocycle and to enhance comprehension of the physiological mecanisms involved in the lower O2 consumption observed.

DETAILED DESCRIPTION:
The training program proposed in this study is realised on an handmade ergocycle which allows almost pur eccentric contractions.

Fifteen healthy volunteers realize a incremental test until exertion on a concentric ergometer. If the minimal power output of 200W is reached, the volunteers are familiarized with eccentric exercise during several bouts of exercise. This habituation session allows avoiding the secondary muscular effects of high intensity eccentric exercise.

Then, volunteers could take part in a two-stepped eccentric protocol: 1) an incremental test consisting in 3 stages. Each stage lasts 4 minutes.

2) A constant-load test realized at 320W during 6 minutes. Each test is realized twice: at 50 and 80 rpm and sequence is randomly assigned.

[One step (incremental or constant load) = two tests (50 and 80 rpm)]

During each step, oxygen consumption is continuously measured, as well as cardiac output and muscular activity and intramuscular oxygen kinetic.

ELIGIBILITY:
Inclusion Criteria:

* - Males
* IMC <30
* physically active
* Pmax concentric > 200W
* Pmax > Pmax théo sédentaire

Exclusion Criteria:

* cardio pulmonary, osteo articulary or muscular diseases
* Eccentric based physical activities or sports (weight liftering, alpine skiing)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption (VO2 ml/min) | at day 1
  Oxygen consumption (VO2) is continuously assesse during exercises at 50 and 80 rpm.

SECONDARY OUTCOMES:
Cardiac output( l/min) | at day 1
muscular oxygen kinetic (arbitrary unit and %) | at day 1
Muscular activity (mV) | at day 1 during one and half minute (1min30s)
  Muscular activity is measured during one and half minute, at the end of each stage
VO2 (ml/min) | at day 1
  VO2 is continously assessed during the constant-load exercise

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France